CLINICAL TRIAL: NCT03914365
Title: Randomized Controlled Trial Comparing Ultrasound-guided Pudendal Nerve Block to Ultrasound-guided Penile Nerve Block for Analgesia Following Pediatric Circumcision
Brief Title: Pudendal Nerve Block vs Penile Nerve Block for Analgesia During Pediatric Circumcision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Katherine Moore, Md FRCSC Pediatric Urologist, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-4132
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Male Circumcision; Regional Anesthesia
Keywords: Circumcision; Penile block; Pudendal block; Pediatric

STUDY DESIGN:
Intervention Model Description: Randomized blinded parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Five regional anesthesia experienced anesthesiologists not involved in the subsequent intraoperative or postoperative care of the patient will perform blocks. Pain scores using the FLACC score(16) will be recorded in the PACU and ambulatory step down unit at 5, 30, 60 and 120 minutes postoperatively by trained and blinded nurses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-guided pudendal nerve block (PNB) (Active Comparator): Standard circumcision under general anaesthesia with ultrasound-guided pudendal nerve block.Pudendal nerve block patients will be positioned dorsally with the legs in the " frog " position (hips in abduction, knees flexed, sole of the feet together). An ultrasound-guided technique will be used as described previously. A linear probe will be positioned horizontally between the ischiatic tuberosity and the rectum. The ischiorectal fossa is then located between these two landmarks. Using a sterile tech-nique, an echogenic 22 gauge, 50 mm block needle will be inserted out of plane on the superior edge of the probe, midline between the ischiatic tuberosity and the rectum. After feeling two distinct fascial " clics " and confirmation of correct needle posi-tioning in the ischiorectal fossa under ultrasound, 0,2 mL/kg (max 10mL) of ropiva-caine 0,25% will be injected under real-time ultrasound-guidance after negative aspiration. The same technique will be repeated on the contralateral side.
  Interventions: Procedure: Ultrasound-guided pudendal nerve block (PNB) and Ultrasound-guided penile nerve block (DPNB)
- Ultrasound-guided penile nerve block (DPNB) (Active Comparator): Standard circumcision under general anaes-thesia with ultrasound-guided penile nerve block.Penile nerve block patients will be positioned in the supine position. An ultrasound-guided technique will be used as described previously. A linear probe will be placed transversely at the base of the penis while an assistant applies caudal traction to the penis. The penile neurovascular sheath is then located just above the corpus cavernosum. The dorsal penile nerve, dorsal penile artery and penile deep dorsal vein are visualized deep to Buck's fascia. Using a sterile technique, a 25 gauge, 1,5 inch needle will be inserted in-plane from lateral to medial so that the needle tip is placed into the penile neurovascular sheath, 0,1 mL/kg (max 4 mL) of ropivacaine 0,25% will be injected under real-time ultrasound guidance while retracting the needle so that the local anaesthetic solution spreads bilaterally filling the neurovascular space.
  Interventions: Procedure: Ultrasound-guided pudendal nerve block (PNB) and Ultrasound-guided penile nerve block (DPNB)

INTERVENTIONS:
Procedure: Ultrasound-guided pudendal nerve block (PNB) and Ultrasound-guided penile nerve block (DPNB) — Our primary objective is to compare analgesia between the two blocks during and after pediatric circumcisions to minimize post-operative pain.

SUMMARY:
Pediatric circumcision has been realized since the beginning of human civilization. In the United States, a 2014 review revealed a 81% prevalence of men 14-59 years old being circumcised.

Circumcision surgery is mostly performed on an ambulatory basis. The best analgesia technique for this procedure has yet to be determined. Local, regional, general anaesthesia or even combinations have been described. The Dorsal Penile Nerve Block (DPNB) has been shown to be superior to topical analgesia in neonatal circumcision. A 2008 Cochrane review showed no difference in pain scores between caudal block and DPNB, but described more motor block with caudal block. For this reason, the 2017 Canadian Urological Association guidelines review recommends using DPNB with a ring block as a standard of care for neonatal circumcision with-out general anaesthesia. However, DPNB does not provide reliable coverage of the ventral surface of the penis and frenulum. Pudendal nerve block (PNB) is another regional anaesthesia technique gaining in popularity with the now widespread use of ultrasound guidance. However, it is still unclear if PNB can give better outcomes than DPNB. The ultrasound-guided pudendal nerve block has only been recently described and was not reviewed as an option at the time of the guidelines writing.

PNB can be performed using surface landmarks, with nerve stimulation or with ultra-sound-guidance. It has already been proven to have lower surgical complication rates than caudal block for hypospadias surgeries. Regarding DPNB, a variety of techniques have been described using either surface landmarks or ultrasound guidance. In the past ten years, two RCTs in Lebanon and Turkey compared PNB and DPNB for penile surgeries, showing lower pain scores and lower narcotics consumption in the pudendal nerve block group. None of these studies used ultrasound-guidance.

The investigators perform more than a hundred pediatric circumcisions yearly for medical indications. The surgery is done under general anaesthesia in association with either PNB or DPNB, depending on the anesthesiologist's preference. The primary objective is to compare analgesia between the two blocks during and after pediatric circumcisions to minimize post-operative pain. The research team will compare peri and postoperative pain in children receiving either ultrasound-guided pudendal nerve block or ultrasound-guided dorsal penile nerve block for circumcision surgery.

DETAILED DESCRIPTION:
All patients will receive inhalational anaesthesia induction with a mixture of oxygen/nitrous oxide and 6% sevoflurane. Nitrous oxide will be discontinued after loss of consciousness. Standard monitoring will be applied including electrocardiography, pulse oxymetry, capnography and non-invasive blood pressure monitoring. After establishing intravenous access, anaesthesia will be deepened using propofol 1 to 3 mg/kg and fentanyl 1 mcg/kg before laryngeal mask airway insertion or intubation. Neuromuscular blockade will not be administered. Maintenance of anaesthesia will be provided with sevoflurane with an end tidal sevoflurane between 1 and 1,5 MAC.

Five regional anesthesia experienced anesthesiologists not involved in the subsequent intraoperative or postoperative care of the patient will perform blocks.

Pudendal nerve block patients will be positioned dorsally with the legs in the " frog " position (hips in abduction, knees flexed and sole of the feet together). An ultrasound-guided technique will be used as described previously. A linear probe will be positioned horizontally between the ischiatic tuberosity and the rectum. The ischiorectal fossa is then located between these two landmarks. Using a sterile technique, an echogenic 22 gauge, 50 mm block needle will be inserted out of plane on the superior edge of the probe, midline between the ischiatic tuberosity and the rectum. After feeling two distinct fascial " clics " and confirmation of correct needle positioning in the ischiorectal fossa under ultrasound, 0,2 mL/kg (max 10mL) of ropivacaine 0,25% will be injected under real-time ultrasound-guidance after negative aspiration. The same technique will be repeated on the contralateral side.

Penile nerve block patients will be positioned in the supine position. An ultrasound-guided technique will be used as described previously. A linear probe will be placed transversely at the base of the penis while an assistant applies caudal traction to the penis. The penile neurovascular sheath is then located just above the corpus cavernosum. The dorsal penile nerve, dorsal penile artery and penile deep dorsal vein are visualized deep to Buck's fascia. Using a sterile technique, a 25 gauge, 1,5 inch needle will be inserted in-plane from lateral to medial so that the needle tip is placed into the penile neurovascular sheath, 0,1 mL/kg (max 4 mL) of ropivacaine 0,25% will be injected under real-time ultrasound guidance while retracting the needle so that the local anaesthetic solution spreads bilaterally filling the neurovascular space.

The heart rate and blood pressure will be recorded before the block and every 5 minutes after block completion by the anaesthesiologist unaware of block assignment involved in the intraoperative and postoperative care of the patient. Surgical incision will be delayed for a minimum of 15 minutes after block completion. Three surgeons will perform all circumcisions using the same surgical technique. Any in-crease in blood pressure or heart rate of more than 20% above baseline within 20 minutes of block completion will be treated with an additional propofol bolus (1mg/kg) or by increasing end-tidal sevoflurane to allow for onset of the block. Any increase in blood pressure or heart rate of more than 20% above baseline 20 minutes or more after the block will be considered inadequate analgesia and will be supplemented with fentanyl 1 mcg/kg. All patients will receive dexamethasone 0,1 mg/kg (max 8 mg) and ondansetron 0,1 mg/kg (max 4 mg). Ketorolac 0,5 mg/kg (max 30 mg) will also be administered at the end of the surgery.

Pain scores using the FLACC score(16) will be recorded in the post-anesthesia care unit (PACU) and ambulatory step down unit at 5, 30, 60 and 120 minutes postoperatively by trained and blinded nurses. A pain score of 4 or higher in the PACU will lead to analgesic administration. A first dose of nalbuphine 0,1 mg/kg will be administered. If inadequate, incremental doses of morphine 0,05 mg/kg will be given until adequate analgesia is achieved. Pain will also be evaluated by parents at home using the parent postoperative pain measure (PPPM) scale at 6, 12 and 24 hours postoperatively. The parents will be instructed by a trained nurse on how to assess the child's pain using this pain measure. Patients will be prescribed acetaminophen 15 mg/kg q 4h regularly (maximum 5 doses/24 hours), ibuprofen 10 mg/kg q 8h regularly and morphine 0,1 mg/kg q 4h as needed.

ELIGIBILITY:
Inclusion Criteria:

* Male 1-12 yo undergoing elective circumcision for medical reasons

Exclusion Criteria:

* Allergy to local anaesthetics or medication used in the study Coagulopathy Infection at the injection site Neurologic or neuromuscular disease ASA classification ≥ 4

Ages: 1 Year to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Impact of regional block on FLACC pain scores after circumcision | 24 hours
  Impact of regional block on pain scores (FLACC score) during the 24 h post-operative period: at 5-30-60-120 minutes postoperative in hospital. The FLACC score (The Face, Legs, Activity, Cry, Consolability scale) The scale is scored in a range of 0-10 with 0 representing no pain. Will be used in the hospital at 5-30-60 and 120 minutes postop.
Impact of regional block on PPPM pain scores after circumcision | 24 hours
  Impact of regional block on PPPM pain scores (parent's postoperative pain measure) during the 24 h post-operative period at 6-12-24h postop at home.
  PPPM score (parents' postoperative pain measure). The scale is scored in a range of 0-15 with 0 representing no pain. Scores 6 and higher represent significant pain. Will be used at home at 6-12-and 24h postop.

SECONDARY OUTCOMES:
Impact of regional block on analgesic consumption after circumcision | 24 hours
  Impact of regional block on analgesic consumption during the first 24h post-operative period.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dave S, Afshar K, Braga LH, Anderson P. Canadian Urological Association guideline on the care of the normal foreskin and neonatal circumcision in Canadian infants (full version). Can Urol Assoc J. 2018 Feb;12(2):E76-E99. doi: 10.5489/cuaj.5033. Epub 2017 Dec 1. No abstract available. PMID 29381458
- [Background] Morris BJ, Bailis SA, Wiswell TE. Circumcision rates in the United States: rising or falling? What effect might the new affirmative pediatric policy statement have? Mayo Clin Proc. 2014 May;89(5):677-86. doi: 10.1016/j.mayocp.2014.01.001. Epub 2014 Apr 2. PMID 24702735
- [Background] Sorokan ST, Finlay JC, Jefferies AL; Canadian Paediatric Society, Fetus and Newborn Committee, Infectious Diseases and Immunization Committee. Newborn male circumcision. Paediatr Child Health. 2015 Aug-Sep;20(6):311-20. doi: 10.1093/pch/20.6.311. PMID 26435672
- [Background] Brady-Fryer B, Wiebe N, Lander JA. Pain relief for neonatal circumcision. Cochrane Database Syst Rev. 2004 Oct 18;2004(4):CD004217. doi: 10.1002/14651858.CD004217.pub2. PMID 15495086
- [Background] Howard CR, Howard FM, Fortune K, Generelli P, Zolnoun D, tenHoopen C, deBlieck E. A randomized, controlled trial of a eutectic mixture of local anesthetic cream (lidocaine and prilocaine) versus penile nerve block for pain relief during circumcision. Am J Obstet Gynecol. 1999 Dec;181(6):1506-11. doi: 10.1016/s0002-9378(99)70397-2. PMID 10601936
- [Background] Cyna AM, Middleton P. Caudal epidural block versus other methods of postoperative pain relief for circumcision in boys. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD003005. doi: 10.1002/14651858.CD003005.pub2. PMID 18843636
- [Background] Kendigelen P, Tutuncu AC, Emre S, Altindas F, Kaya G. Pudendal Versus Caudal Block in Children Undergoing Hypospadias Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):610-5. doi: 10.1097/AAP.0000000000000447. PMID 27501015
- [Background] Hecht S, Pineda J, Bayne A. Ultrasound-guided Pudendal Block Is a Viable Alternative to Caudal Block for Hypospadias Surgery: A Single-Surgeon Pilot Study. Urology. 2018 Mar;113:192-196. doi: 10.1016/j.urology.2017.11.006. Epub 2017 Nov 16. PMID 29155191
- [Background] Tutuncu AC, Kendigelen P, Ashyyeralyeva G, Altintas F, Emre S, Ozcan R, Kaya G. Pudendal Nerve Block Versus Penile Nerve Block in Children Undergoing Circumcision. Urol J. 2018 May 3;15(3):109-115. doi: 10.22037/uj.v0i0.4292. PMID 29299888
- [Background] Naja Z, Al-Tannir MA, Faysal W, Daoud N, Ziade F, El-Rajab M. A comparison of pudendal block vs dorsal penile nerve block for circumcision in children: a randomised controlled trial. Anaesthesia. 2011 Sep;66(9):802-7. doi: 10.1111/j.1365-2044.2011.06753.x. Epub 2011 Jul 25. PMID 21790518
- [Background] Gaudet-Ferrand I, De La Arena P, Bringuier S, Raux O, Hertz L, Kalfa N, Sola C, Dadure C. Ultrasound-guided pudendal nerve block in children: A new technique of ultrasound-guided transperineal approach. Paediatr Anaesth. 2018 Jan;28(1):53-58. doi: 10.1111/pan.13286. Epub 2017 Dec 5. PMID 29205687
- [Background] Suleman MI, Akbar Ali AN, Kanarek V, Li M, Patel A. Ultrasound Guided In-Plane Penile Nerve Block for Circumcision: A New, Modified Technique Suggests Lower Anesthetic Volume and Narcotic Use. Middle East J Anaesthesiol. 2016 Oct;23(6):647-53. PMID 29939703
- [Background] McGrath PJ, Walco GA, Turk DC, Dworkin RH, Brown MT, Davidson K, Eccleston C, Finley GA, Goldschneider K, Haverkos L, Hertz SH, Ljungman G, Palermo T, Rappaport BA, Rhodes T, Schechter N, Scott J, Sethna N, Svensson OK, Stinson J, von Baeyer CL, Walker L, Weisman S, White RE, Zajicek A, Zeltzer L; PedIMMPACT. Core outcome domains and measures for pediatric acute and chronic/recurrent pain clinical trials: PedIMMPACT recommendations. J Pain. 2008 Sep;9(9):771-83. doi: 10.1016/j.jpain.2008.04.007. Epub 2008 Jun 17. PMID 18562251
- [Background] Boric K, Jelicic Kadic A, Boric M, Zarandi-Nowroozi M, Jakus D, Cavar M, Dosenovic S, Jeric M, Batinic M, Vukovic I, Puljak L. Outcome domains and pain outcome measures in randomized controlled trials of interventions for postoperative pain in children and adolescents. Eur J Pain. 2019 Feb;23(2):389-396. doi: 10.1002/ejp.1313. Epub 2018 Sep 21. PMID 30179284
- [Background] Berde CB, Walco GA, Krane EJ, Anand KJ, Aranda JV, Craig KD, Dampier CD, Finkel JC, Grabois M, Johnston C, Lantos J, Lebel A, Maxwell LG, McGrath P, Oberlander TF, Schanberg LE, Stevens B, Taddio A, von Baeyer CL, Yaster M, Zempsky WT. Pediatric analgesic clinical trial designs, measures, and extrapolation: report of an FDA scientific workshop. Pediatrics. 2012 Feb;129(2):354-64. doi: 10.1542/peds.2010-3591. Epub 2012 Jan 16. PMID 22250028
- [Background] Chambers CT, Reid GJ, McGrath PJ, Finley GA. Development and preliminary validation of a postoperative pain measure for parents. Pain. 1996 Dec;68(2-3):307-13. doi: 10.1016/s0304-3959(96)03209-5. PMID 9121819
- [Background] Manworren RC, Hynan LS. Clinical validation of FLACC: preverbal patient pain scale. Pediatr Nurs. 2003 Mar-Apr;29(2):140-6. PMID 12723828
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Nilsson S, Finnstrom B, Kokinsky E. The FLACC behavioral scale for procedural pain assessment in children aged 5-16 years. Paediatr Anaesth. 2008 Aug;18(8):767-74. doi: 10.1111/j.1460-9592.2008.02655.x. PMID 18613934
- [Background] Willis MH, Merkel SI, Voepel-Lewis T, Malviya S. FLACC Behavioral Pain Assessment Scale: a comparison with the child's self-report. Pediatr Nurs. 2003 May-Jun;29(3):195-8. PMID 12836995
- [Derived] Boisvert-Moreau F, Turcotte B, Albert N, Singbo N, Moore K, Boivin A. Randomized controlled trial (RCT) comparing ultrasound-guided pudendal nerve block with ultrasound-guided penile nerve block for analgesia during pediatric circumcision. Reg Anesth Pain Med. 2023 Mar;48(3):127-133. doi: 10.1136/rapm-2022-103785. Epub 2022 Nov 17. PMID 36396298